CLINICAL TRIAL: NCT00775671
Title: Comparative Effect of Nebivolol vs. Metoprolol on Insulin Sensitivity and Fibrinolytic Balance in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 080496
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Nebivolol 5mg by mouth daily for 12 weeks.
  Interventions: Drug: placebo; Drug: Nebivolol
- Metoprolol (Active Comparator): Metoprolol ER 100mg by mouth daily for 12 weeks.
  Interventions: Drug: placebo; Drug: Metoprolol

INTERVENTIONS:
Drug: placebo — Placebo pill by mouth daily for 21 days followed by either Nebivolol 5 mg by mouth daily or metoprolol ER 100mg by mouth daily for 12 weeks.
Drug: Nebivolol — Nebivolol 5 mg by mouth daily for 12 weeks.
  Arms: Nebivolol
Drug: Metoprolol — Metoprolol ER 100mg by mouth daily for 12 weeks.
  Arms: Metoprolol

SUMMARY:
Test the hypothesis that nebivolol treatment improves fibrinolytic balance and insulin sensitivity compared to metoprolol treatment in individuals with metabolic syndrome.

DETAILED DESCRIPTION:
1. Test the hypothesis that nebivolol treatment decreases PAI-1 antigen and activity and improves fibrinolytic balance compared to metoprolol treatment in individuals with metabolic syndrome.
2. Test the hypothesis that nebivolol treatment improves insulin sensitivity compared to metoprolol treatment in individuals with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects, 18 to 70 years of age, inclusive
2. For female subjects, the following conditions must be met:

   * postmenopausal status for at least 1 year, or
   * status-post surgical sterilization, or
   * if of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-hcg testing prior to drug treatment and on every study day
3. Metabolic syndrome as defined by 3 or more of the following:

   * Fasting plasma glucose of at least 100 mg/dL (5.5 mmol/L)
   * Serum triglycerides of at least 150 mg/dL (1.7 mmol/L)
   * Serum HDL cholesterol less than 40 mg/dL (1.04 mmol/L) in men and 50 mg/dL in women
   * Blood pressure of at least 130/85 mmHg
   * Waist girth of more than 102 cm in men or 88 cm in women

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Diabetes type 1 or type 2, as defined by a fasting glucose of 126 mg/dL or greater or the use of anti-diabetic medication
2. Use of hormone replacement therapy
3. Change in statin therapy within the last 6 months
4. In hypertensive subjects, a seated systolic blood pressure greater than 179 mmHg or a seated diastolic blood pressure greater than 110 mmHg
5. Pregnancy
6. Breast-feeding
7. Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second- or third-degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
8. Treatment with anticoagulants
9. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
10. History or presence of immunological or hematological disorders
11. Diagnosis of asthma
12. Clinically significant gastrointestinal impairment that could interfere with drug absorption
13. Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >2.0 x upper limit of normal range)
14. Impaired renal function (serum creatinine >1.5 mg/dl)
15. Hematocrit <35%
16. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
17. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
18. Treatment with lithium salts
19. History of alcohol or drug abuse
20. Treatment with any investigational drug in the 1 month preceding the study
21. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
22. Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
23. Inability to swallow capsules

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Ayers K, Byrne LM, DeMatteo A, Brown NJ. Differential effects of nebivolol and metoprolol on insulin sensitivity and plasminogen activator inhibitor in the metabolic syndrome. Hypertension. 2012 Apr;59(4):893-8. doi: 10.1161/HYPERTENSIONAHA.111.189589. Epub 2012 Feb 21. PMID 22353614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants answered recruitment advertisments. All qualifying participants had Metabolic Syndrome.
Pre-assignment Details: Participants that met inclusion criteria stopped their antihypertensive medications for 3 weeks before study start. All participants took a placebo pill daily for 21 days and had baseline measurements done.
Groups:
- Metoprolol: Metoprolol ER 100mg by motuh daily for 12 weeks.
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.5) | 47.4 (8.5) | 44.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Secondary Outcome: Measurement of Insulin Sensitivity
Description: The change in insulin sensitivity index, from baseline to after 12 weeks of treatment. Calculated from the intravenous glucose tolerance test at baseline and at 12 weeks.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: 10-4xmin-1 per mU/L
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 23 | 23
10-4xmin-1 per mU/L | 0.04 (2.19) | -1.5 (2.5)

2. Primary Outcome: Marker of Fibrinolysis
Description: Concentration of plasminogen activator inhibitor 1 (PAI-1)antigen.
Time Frame: After 12 weeks of study drug
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nebivolol | Metoprolol
Number analyzed (Participants) | 23 | 23
ng/mL | 10.5 (6.2) | 12.3 (7.8)

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: Time from washing off antihypertensive medication, taking placebo for 21 days, and taking study drug for 12 weeks.
Arm/Group | Nebivolol | Metoprolol
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 14/23 | 7/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol (N=23) | Metoprolol (N=23)
congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
Headache (General disorders) | 3 (3) | 1 (1)
Sore Throat (General disorders) | 2 (2) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2)
palpitations (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes